CLINICAL TRIAL: NCT01990183
Title: CareToy - A Modular Smart System for Infants' Rehabilitation at Home Based on Mechatronic Toys
Acronym: CareToy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Fondazione Stella Maris (Other)
Collaborators: BioRobotics Institute (Other); STMicroelectronics SRL, Italy (Unknown); University of Ljubljana (Other); University of Hamburg-Eppendorf (Other); Fonden for Helen Elsass Center, Denmark (Unknown); Marketing Research & Development SPA, Italy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICT-2011.5.1-287932
Record Dates: First submitted 2013-11-07; First posted 2013-11-21 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Preterms at Risk for Developmental Disorders
Keywords: preterm infants; early intervention; enrichment; cognitive, motor, visual development; tele-rehabilitation
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CareToy (Experimental): CareToy intervention
  Interventions: Device: CareToy
- Standard Care (Other): Standard Care
  Interventions: Other: Standard Care

INTERVENTIONS:
Device: CareToy — Infants randomized in the Intervention Group will begin the habilitation intervention immediately after evaluation at baseline. Rehabilitation staff, in accordance with each infant's needs and clinical characteristics, will set up the CareToy System to perform individualized intervention packages and its user's manual. So a personalized CareToy System will be delivered at infant's home. Moreover parents will attend a training course to use it. During each daily home - session (about 30 - 45 minutes overall) it will be proposed to the child various interactive activities in supine, prone and sitting position. The intervention phase lasts 4 weeks and each session will be remotely monitored by the rehabilitation staff.
  Arms: CareToy
Other: Standard Care — Current care advices in the management of preterm infants in the first months of life
  Arms: Standard Care

SUMMARY:
Stroke and other neurological conditions affect the population of infants in percentages that cannot be considered marginal. Preterm infants are the highest infants at risk for neurological damage. Currently, infants have rehabilitation sessions few times a week in rehabilitation centres but according to basic neuroscience it would be necessary to provide them with an early, intensive and multiaxial intervention. One option to reduce the cost of the entire European Healthcare System while increasing the practice of rehabilitation is to devise therapies and technologies that can be administered at home by caregivers and telemonitored by rehabilitation staff. The aim of this proposal is to promote early intervention in the first year of life and to reinforce therapy by "CareToy": a portable low cost smart system telemonitored thus augmenting the clinical effectiveness of the therapy while reducing the cost. The smart system is based on a common baby gym, composed of different modules: a) an instrumented baby gym with mechatronic hanging toys, so that the infants' actions on the gym can be measured and stimulated, b) a vision module, for measuring and promoting infants' attention and gaze movements and c) a sensorized mat for measuring and promoting postural control. Each module will also incorporate built-in signal processor, memory and wireless communication. A fourth telerehabilitation module completes the system that allows the system to remotely communicate with the rehabilitation staff for monitoring and assessing the rehabilitation techniques. CareToy and the effectiveness of home rehabilitation based on this system will be validated by clinical trials on at least 50 preterm infants. The result of this project could have a large impact. CareToy may become a commercial product, manufactured on a large scale and distributed not only in rehabilitation centres but also at homes, sold or rented by the Health Care System to families as a therapeutic tool for care intensity.

DETAILED DESCRIPTION:
Study population will be made up of premature infants recruited at the local Department of Neonatology. The eligibility of infants, i.e. children who meet the criteria for inclusion and exclusion, will be evaluated by the Neonatology team. Recruitment should take place after discharge from Neonatal Intensive Care Unit (NICU) until the age stated by inclusion criteria and will begin with the signing of the participation agreement by the parents. During the recruitment extensive perinatal data will be collected from medical records. Each clinical centre will maintain these data in an internal database storing. Every child will be evaluated on the basis of a standard neurological examination supplemented by movement analysis on video recording using Prechtl's Method Qualitative Assessment of General Movements.

The sample will be randomized in two groups in order to compare the effectiveness of the CareToy intervention program vs standard care on motor, cognitive and visual development. We designed the study as randomized clinical trial. The sample size was calculated on the basis of the primary outcome measure (Infant Motor Profile [IMP], see Outcome measures).

Before the starting of the RCT we have planned a short pilot phase where few infants in order to assess the feasibility of the CareToy training and to tune and set-up the CareToy system and the rehabilitation packages. These cases will follow the same steps planned for the RCT.

ELIGIBILITY:
Inclusion Criteria:

* gestational age ≥ 28+0 weeks and 32+6 weeks
* corrected age at baseline: between 3 and 9 months;
* achievement of predefined cut off scores in gross motor ability derived from Ages & Stages Questionnaire® Third Edition (ASQ-3), in relation to corrected age (Bricker and Squires, 1999)

In detail:

* 4 months form (from 3 months to 4 months 30 days) score ≥ 10;
* 6 months form (from 5 months to 6 months 30 days) score ≥ 5 - < 50;
* 8 months form (from 7 months to 8 months 30 days) ≥ 10 - <30

Exclusion Criteria:

* infants with gestational age < 28 weeks or ≥ 33 weeks
* infants small for gestational age (i.e. weight below the 10th, ref)
* presence of brain damage (i.e. brain malformation, intra-ventricular haemorrhage [IVH] >1 ; any degree of periventricular leukomalacia (ref)
* known epilepsy or other form of seizure
* severe sensory deficits (blindness, deafness)
* other severe non neurological malformations
* participation in other experimental studies having rehabilitation aims

Ages: 3 Months to 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2013-07; Primary Completion 2015-04 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Changes on Infant Motor Profile (IMP) | T0(baseline, 1week before beginning of Study period);T1 (within 1 week after the end of the first training/control period; before the cross-over); T2 (within 1 week after the end of the second training/control 2nd period, after cross-over), T3: 18 months
  IMP is a reliable video-based assessment of motor behaviour in infancy from 3 to 18 months. It addresses to the child's motor abilities and evaluates motor behaviour in five domains: (1) variation, (2) variability (ability to select motor strategies), (3) movement fluency, (4) movement symmetry, and (5) motor performance. It has been validated in preterm and full term infants. This tool is intended to detect and quantify changes after intervention and it is reported as having a satisfactory intra and inter observer reliability and a very good concurrent validity with Alberta Infant Motor Scale and Touwen Infant Neurological Examination.

SECONDARY OUTCOMES:
Changes on Alberta Infant Motor Scale (AIMS) | T0 (baseline,1wk before beginning of Study period);T1(within 1 wk after end of 1st training/control period; before cross-over);T2 (within 1wk after end of 2nd training/control 2nd period, after cross-over) T3 (18 mths of corrected age)
  This scale examines delayed and abnormal motor development in infants overtime and is valid for assessment from term until 18 months of age. It has a good psychometric properties, it is quick to administer with limited handling and focuses on achievement of motor milestones, quality of posture and movement outcomes. Sensitivity of AIMS items has been demonstrated in differentiate preterm's infant motor development, that typically results in lower scores, and full term infants motor development.
CareToy for Clinics (CareToy C) | T0 (baseline, 1week before beginning of Study period);T1 (within 1 week after the end of the first training/control period; before the cross-over); T2 (within 1 week after the end of the second training/control 2nd period, after cross-over)
  CareToy Evaluation Packages will be carried out using a highly equipped system, called Caretoy C in a subgroup of the enrolled infants. This evaluation is mainly composed by visual packages designed to evaluate some different infants visual abilities i.e. attention, audio-visual, fixation shift and novelty.
Changes on Teller Acuity Cards | T0 (baseline,1wk before beginning of Study period);T1(within 1 wk after end of 1st training/control period; before cross-over);T2 (within 1wk after end of 2nd training/control 2nd period, after cross-over) T3 (18 mths of corrected age)
  Teller Acuity Cards II is a paediatric test used to evaluate visual acuity. It is based on behavioural response by judging infant's attention to a series of cards showing stripes of different widths. This tool allows rapid assessment of resolution (grating) visual acuity in infants, young children, and other populations where verbal response to recognition (letter) visual acuity charts is difficult or impossible. It evaluates infants' acuity development and it has been used in several studies for diagnostic purposes and to measure results of early intervention.
Changes on Bayley III - Cognitive subscale | T0 (baseline, 1week before beginning of Study period);T3: 18 months of Corrected Age (CA)
  his scale is sensitive in detecting differences between normative sample and children at risk for delayed development, such as premature infants. It has normative value referenced assessments, with means of 100 and Standard Deviation [SD] of 15 points. Children whose scores are 2 SDs below the normative value in a domain are considered as having a significant delay in that domain. Bayley---III is appropriate for administration to children between the ages of 1 month and 42 months (although norms extend downward to age 16 days). The Bayley III revision includes Cognitive, Language, Motor, Social-Emotional, and Adaptive Behaviour scales. Items on the cognitive subscale assess sensor-motor development, exploration, manipulation, object relatedness, concept formation, problem-solving and memory, all functions promoted during the CareToy sessions.

OTHER OUTCOMES:
Ages & Stages Questionnaire (ASQ) | T0 (baseline,1wk before beginning of Study period);T1(within 1 wk after end of 1st training/control period; before cross-over);T2 (within 1wk after end of 2nd training/control 2nd period, after cross-over); T3 (18 mths of corrected age)
  It has been developed as a screening tool for developmental delay in infants in numerous paediatric populations with reported sensitivity, a measure of true positives, and specificity, a measure of true negatives, varying, with most studies reporting higher accuracy in at - risk populations.
  This questionnaire will be given to parents after enrolment in order to define the most appropriate starting time for each infant.
Social - Emotional Scale of BSID-III | T0 (baseline,1wk before beginning of Study period);T1(within 1 wk after end of 1st training/control period; before cross-over);T2 (within 1wk after end of 2nd training/control 2nd period, after cross-over); T3 (18 mths of corrected age)
  The survey uses this observational rating scale that provides a general indication of the infant's level of social- emotional development and information about whether or not sensory processing difficulties are present.
Parenting Stress Index (PSI) | T0 (baseline,1wk before beginning of Study period);T1(within 1 wk after end of 1st training/control period; before cross-over);T2 (within 1wk after end of 2nd training/control 2nd period, after cross-over) T3 (18 mths of corrected age)
  This is a self-report questionnaire designed to identify specific parental, child, and situational characteristics most commonly associated with dysfunctional parenting. Currently, the PSI is mostly used as a screening instrument for early identification of parent- child systems, which are under stress and at risk of developing dysfunctional parenting behaviour. Validity of PSI is good and has been established in numerous studies on children with developmental problems, behaviour problems, disabilities and illnesses, as well as studies of at- risk families, and cross - cultural studies

CONTACTS AND LOCATIONS:
Locations (2):
- Helene Elsass Center, Holmegaardsvej 28, Charlottenlund, Denmark
- IRCCS Stella Maris Foundation, Calambrone, Pisa, Italy

REFERENCES:
- [Derived] Rizzi R, Menici V, Cioni ML, Cecchi A, Barzacchi V, Beani E, Giampietri M, Cioni G, Sgandurra G; Clinical CareToy-R Consortium. Concurrent and predictive validity of the infant motor profile in infants at risk of neurodevelopmental disorders. BMC Pediatr. 2021 Feb 6;21(1):68. doi: 10.1186/s12887-021-02522-5. PMID 33549070
- [Derived] Sgandurra G, Beani E, Inguaggiato E, Lorentzen J, Nielsen JB, Cioni G. Effects on Parental Stress of Early Home-Based CareToy Intervention in Low-Risk Preterm Infants. Neural Plast. 2019 Jan 22;2019:7517351. doi: 10.1155/2019/7517351. eCollection 2019. PMID 30804992
- [Derived] Sgandurra G, Lorentzen J, Inguaggiato E, Bartalena L, Beani E, Cecchi F, Dario P, Giampietri M, Greisen G, Herskind A, Nielsen JB, Rossi G, Cioni G; CareToy Consortium. A randomized clinical trial in preterm infants on the effects of a home-based early intervention with the 'CareToy System'. PLoS One. 2017 Mar 22;12(3):e0173521. doi: 10.1371/journal.pone.0173521. eCollection 2017. PMID 28328946
- [Derived] Sgandurra G, Bartalena L, Cioni G, Greisen G, Herskind A, Inguaggiato E, Lorentzen J, Nielsen JB, Sicola E; CareToy Consortium. Home-based, early intervention with mechatronic toys for preterm infants at risk of neurodevelopmental disorders (CARETOY): a RCT protocol. BMC Pediatr. 2014 Oct 15;14:268. doi: 10.1186/1471-2431-14-268. PMID 25319764
- See also: Related Info — http://www.caretoy.eu